CLINICAL TRIAL: NCT05276973
Title: Phase I/IB Safety and Pharmacodynamic Study of Neoadjuvant (NACT) Paclitaxel and Carboplatin With Ipatasertib as Initial Therapy of Ovarian Cancer PTMA 100805
Brief Title: Testing the Addition of Ipatasertib to the Usual Chemotherapy Treatment (Paclitaxel and Carboplatin) for Stage III or IV Epithelial Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-01930; NCI-2022-01930 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY027 (Other: NRG Oncology); NRG-GY027 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-03-11; First posted 2022-03-14 (Actual); Results first posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10

CONDITIONS: Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube High Grade Serous Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal High Grade Serous Adenocarcinoma; Stage III Fallopian Tube Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8; Unresectable Fallopian Tube Endometrioid Adenocarcinoma; Unresectable Fallopian Tube High Grade Serous Adenocarcinoma; Unresectable Ovarian Endometrioid Adenocarcinoma; Unresectable Ovarian High Grade Serous Adenocarcinoma; Unresectable Primary Peritoneal Endometrioid Adenocarcinoma; Unresectable Primary Peritoneal High Grade Serous Adenocarcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Biopsy; Carboplatin; ipatasertib; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (paclitaxel, carboplatin, ipatasertib) (Experimental): Patients receive paclitaxel IV at 175mg/m2 over 3 hours and carboplatin IV at AUC 5 over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive ipatasertib PO QD until 24 hours before surgery in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Drug: Carboplatin; Drug: Ipatasertib; Drug: Paclitaxel

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase I/IB trial tests the safety, side effects, and best dose of ipatasertib in combination with paclitaxel and carboplatin in treating patients with stage III or IV epithelial ovarian cancer. Ipatasertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Paclitaxel is in a class of medications called taxanes. It stops tumor cells from growing and dividing and may kill them. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Giving ipatasertib in combination with paclitaxel and carboplatin may lower the chance of the tumor growing or spreading for longer than the paclitaxel and carboplatin alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and the dose limiting toxicities (DLTs) of ipatasertib in combination with paclitaxel and carboplatin as neoadjuvant chemotherapy for ovarian cancer.

II. To determine the feasibility of the treatment regimen once the MTD is estimated.

III. To assess the toxicities of ipatasertib in combination with paclitaxel and carboplatin by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OBJECTIVE:

I. Objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 prior to interval debulking surgery (IDS).

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To evaluate the change of phosphorylated (p)PRAS40 expression in the pre-treatment tumor versus (vs.) on-treatment tumor.

II. To identify the pharmacokinetics of ipatasertib in the tissue and blood. III. To correlate antitumor response with genomic alterations in PI3K pathway genes (PTEN, PIK3CA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1).

IV. To correlate antitumor response with transcriptomic alterations in PI3K pathway genes (PTEN, PIK3CA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1).

V. To correlate response with PTEN loss.

OUTLINE: This is a dose-escalation study of ipatasertib followed by a dose-expansion study.

Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive ipatasertib orally (PO) once daily (QD) until 24 hours before surgery in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of ovarian cancer (ovarian cancer = fallopian tube cancer, ovarian cancer, primary peritoneal cancer). Required data element: submission of pathology report. Patients with the following histologic cell types are eligible:

  * High grade serous
  * Endometrioid adenocarcinoma, grade 3 Genomic/genetic testing results will be a data collection element if performed as part of usual care (germline genetic testing, tumor genomic testing, homologous recombination deficiency [HRD] testing). Genetic/genomic testing results should be uploaded if they become available anytime during conduct of the study
* Appropriate stage for study entry defined as stage III or stage IV based on the following diagnostic workup:

  * History/physical examination within 14 days prior to registration
  * Imaging with computed tomography (CT) chest/abdomen/pelvis (C/A/P) within 28 days prior to registration
* Patients must have evaluable disease or measurable disease defined by RECIST version (v) 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by CT or magnetic resonance imaging (MRI). Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Pre-treatment formalin-fixed, paraffin-embedded (FFPE) tumor block collected from laparoscopy (preferred) or five 18G cores by radiology/interventional radiology (acceptable) must be available for submission
* Disease must be considered unresectable via primary debulking surgery and in need of neoadjuvant chemotherapy (NACT) prior to debulking surgery. This assessment of unresectability can be made via imaging or laparoscopic scoring
* No prior therapy directed at ovarian cancer
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 within 14 days prior to registration
* Absolute neutrophil count >= 1,000/mcl (within 14 days prior to registration)
* Platelets >= 100,000/mcl (within 14 days prior to registration)
* Creatinine =< institutional/laboratory upper limit of normal (ULN) or creatinine clearance (CrCL) or estimated glomerular filtration rate (eGFR) of >= 60 mL/min estimated using either the Cockcroft-Gault equation, the Modification of Diet in Renal Disease Study, or as reported in the comprehensive metabolic panel/basic metabolic panel (eGFR) (within 14 days prior to registration)
* Total bilirubin =< 1.5 x ULN (patients with known Gilbert's disease who have bilirubin level =< 3 x ULN may be enrolled) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x ULN (within 14 days prior to registration)
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Women of childbearing potential (WOCBP) must agree to use two forms of birth control (hormonal or barrier method of birth control; abstinence) agree to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 28 days after the last dose of ipatasertib and agreement to refrain from donating eggs during this same period
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information
* Ability to understand and willingness to sign an institutional review board (IRB) approved written informed consent document (or that of legally authorized representative, if applicable)

Exclusion Criteria:

* Prior treatment with agent(s) targeting PI3K/AKT/mTor pathway
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ipatasertib, paclitaxel or carboplatin
* Currently receiving any other investigational agents or has received an investigational agent within 4 weeks of study registration
* Abnormal gastrointestinal function. This includes gastrointestinal (GI) obstruction or bleeding or signs/symptoms thereof within 3 months of study registration
* Patients with a history of abdominal fistula will be considered eligible if the fistula was surgically repaired or has healed, there has been no evidence of fistula for at least 6 months, and patient is deemed to be at low risk of recurrent fistula
* Received prior radiotherapy to any portion of the abdominal cavity or pelvis
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Patients with active infections requiring intravenous antibiotics
* Patients with diabetes either requiring insulin therapy or with a baseline fasting glucose >= 160 mg/dL and/or high glycosylated hemoglobin (HbA1c) (> 8), suggesting poorly controlled diabetes. Fasting is defined as abstaining from food and drink (with the exception of water) for at least 8 hours
* Patients with grade >= 2 uncontrolled or untreated hypercholesterolemia (> 300 mg/dL) or hypertriglyceridemia (> 300 mg/dL) would be an ineligible
* History of or active inflammatory bowel disease (e.g., Crohn's disease and/or ulcerative colitis) or active bowel inflammation (e.g., diverticulitis)
* Lung disease: Pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia)
* Patients with known brain metastases or leptomeningeal disease are not eligible, as prior treatment directed at ovarian cancer is not allowed
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to registration

  * Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Known clinically significant history of liver disease consistent with Child Pugh class B or C, including active viral or other hepatitis, current drug or alcohol abuse, or cirrhosis
* Pregnant women are excluded from this study because ipatasertib is an oral AKT inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ipatasertib, breastfeeding should be discontinued if the mother is treated with ipatasertib. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2026-02-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Fuh, Principal Investigator — NRG Oncology
Locations (8):
- United States (8):
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Augusta University Medical Center, Augusta, Georgia
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NRG-GY027 opened to accrual on June 27, 2022, and closed to accrual on December 20, 2024 with a total of 25 participants enrolled.
Groups:
- Dose Level 1 (DL1) Escalation Cohort; Dose Level 1 (DL1) Dose Expansion-only Cohort: Paclitaxel at 175 mg/m2 was administered intravenously over 3 hours, and carboplatin at AUC 5 was administered intravenously over 30-60 minutes on Day 1 of each 21-day treatment cycle. Treatment was repeated every 21 days for up to 3 cycles, in the absence of disease progression or unacceptable toxicity. Concurrently, ipatasertib was administered orally at a dose of 200 mg once daily and continued until 24 hours prior to surgery, unless disease progression or unacceptable toxicity.
- Dose Level 2 (DL2) Dose Escalation Cohort: Paclitaxel at 175 mg/m2 was administered intravenously over 3 hours, and carboplatin at AUC 5 was administered intravenously over 30-60 minutes on Day 1 of each 21-day treatment cycle. Treatment was repeated every 21 days for up to 3 cycles, in the absence of disease progression or unacceptable toxicity. Concurrently, ipatasertib was administered orally at a dose of 300 mg once daily and continued until 24 hours prior to surgery, unless disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Dose Level 1 (DL1) Escalation Cohort | Dose Level 1 (DL1) Dose Expansion-only Cohort | Dose Level 2 (DL2) Dose Escalation Cohort
Started (Enrolled and eligible.) | 7 | 13 | 5
Completed (DLT-evaluable patients) | 6 | 12 | 5
Not Completed | 1 | 1 | 0
Not completed — Treated and DLT unevaluable | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who received any amount of protocol therapy
Groups:
- DL1 Escalation Cohort: Participants who were enrolled in the dose escalation phase and received any amount of the assigned DL1 therapy.
- DL1 Dose Expansion-only Cohort: Participants who were enrolled in the dose expansion cohort phase only and received any amount of the assigned DL1 therapy.
- DL2 Dose Escalation Cohort: Participants who were enrolled in the dose escalation phase and received any amount of the assigned DL2 therapy.
- Total: Total of all reporting groups
Arm/Group | DL1 Escalation Cohort | DL1 Dose Expansion-only Cohort | DL2 Dose Escalation Cohort | Total
Number analyzed (Participants) | 7 | 13 | 5 | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [47 to 73] | 66 [44 to 82] | 69 [63 to 80] | 66 [44 to 82]
Age, Customized [Count of Participants; unit: Participants]
  40-49 | 1 | 1 | 0 | 2
  50-59 | 2 | 3 | 0 | 5
  60-69 | 2 | 5 | 3 | 10
  70-79 | 2 | 3 | 2 | 7
  80-89 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 5 | 25
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 11 | 4 | 21
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 6 | 8 | 3 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicities (DLTs) During Dose Escalation Phase
Description: The incidence of DLTs was assessed based on the number of participants who experienced at least one dose-limiting toxicity (DLT) during the Dose Escalation phase, which was used to estimate the maximum tolerated dose (MTD). A DLT was defined as any protocol-specified adverse event that was possibly, probably, or definitely related to study drug combination and occurred during the first cycle of neoadjuvant chemotherapy, unless the event was clearly unrelated to the study therapy. Adverse events were assessed and graded according to NCI CTCAE v5.0.
Time Frame: First cycle of 21 days
Population: Participants who received the assigned DL1 protocol therapy or DL2 protocol therapy and were evaluable for DLTs during dose escalation phase.
Measure: Count of Participants; unit: Participants
Groups:
- DL1 Dose Escalation Cohort: Paclitaxel at 175 mg/m2 was administered intravenously over 3 hours, and carboplatin at AUC 5 was administered intravenously over 30-60 minutes on Day 1 of each 21-day treatment cycle. Treatment was repeated every 21 days for up to 3 cycles, in the absence of disease progression or unacceptable toxicity. Concurrently, ipatasertib was administered orally at a dose of 200 mg once daily and continued until 24 hours prior to surgery, unless disease progression or unacceptable toxicity.
- DL2 Dose Escalation Cohort: Paclitaxel at 175 mg/m2 was administered intravenously over 3 hours, and carboplatin at AUC 5 was administered intravenously over 30-60 minutes on Day 1 of each 21-day treatment cycle. Treatment was repeated every 21 days for up to 3 cycles, in the absence of disease progression or unacceptable toxicity. Concurrently, ipatasertib was administered orally at a dose of 300 mg once daily and continued until 24 hours prior to surgery, unless disease progression or unacceptable toxicity.
Arm/Group | DL1 Dose Escalation Cohort | DL2 Dose Escalation Cohort
Number analyzed (Participants) | 6 | 5
Participants | 1 | 2

2. Primary Outcome: Incidence of Dose-limiting Toxicities (DLTs) During Dose Expansion Phase
Description: The incidence of DLTs was assessed based on the number of participants who experienced at least one DLT during the Dose Expansion phase. This assessment was used to evaluate the feasibility of the treatment regimen at the estimated MTD, specially dose level 1. A DLT was defined as any protocol-specified adverse effect that was possibly, probably, or definitely related to study drug combination and occurred during the first cycle of neoadjuvant chemotherapy, unless the event was clearly unrelated to study therapy. Adverse events were assessed and graded according to NCI CTCAE v.5.0.
Time Frame: First cycle of 21 days
Population: Participants who were treated at the identified MTD level (DL1) and evaluable for DLTs. This population consisted of the 6 DLT-evaluable participants from Dose Escalation Phase and additional 12 DLT-evaluable participants from Dose Expansion Phase.
Measure: Count of Participants; unit: Participants
Groups:
- DL1 Dose Expansion Cohort: Paclitaxel at 175 mg/m2 was administered intravenously over 3 hours, and carboplatin at AUC 5 was administered intravenously over 30-60 minutes on Day 1 of each 21-day treatment cycle. Treatment was repeated every 21 days for up to 3 cycles, in the absence of disease progression or unacceptable toxicity. Concurrently, ipatasertib was administered orally at a dose of 200 mg once daily and continued until 24 hours prior to surgery, unless disease progression or unacceptable toxicity.
Arm/Group | DL1 Dose Expansion Cohort
Number analyzed (Participants) | 18
Participants | 2

3. Primary Outcome: Incidence of Grade 3 or Higher Adverse Events (AEs)
Description: The incidence of grade 3 or higher AEs was assessed based on the number of participants who experienced at least one grade 3 or higher adverse event. Adverse events were graded and categorized according to NCI CTCAE v5.0.
Time Frame: During treatment period and up to 90 days after the last dose of ipatasertib. The median duration of study treatment was 68 days with a range from 1 day to 90 days.
Population: Participants who received any amount of protocol therapy.
Measure: Count of Participants; unit: Participants
Groups:
- DL1 Dose Expansion-only Cohort: Paclitaxel at 175 mg/m2 was administered intravenously over 3 hours, and carboplatin at AUC 5 was administered intravenously over 30-60 minutes on Day 1 of each 21-day treatment cycle. Treatment was repeated every 21 days for up to 3 cycles, in the absence of disease progression or unacceptable toxicity. Concurrently, ipatasertib was administered orally at a dose of 200 mg once daily and continued until 24 hours prior to surgery, unless disease progression or unacceptable toxicity.
Arm/Group | DL1 Dose Escalation Cohort | DL1 Dose Expansion-only Cohort | DL2 Dose Escalation Cohort
Number analyzed (Participants) | 7 | 13 | 5
Participants | 2 | 8 | 5

4. Secondary Outcome: Tumor Response
Description: Tumor response was assessed by RECIST 1.1 at 3 weeks (+/- 7 days) post Cycle 3 of the study treatment and prior to interval debulking surgery (IDS), and it could be repeated any other time if clinically indicated based on symptoms or physical signs suggestive of new or progressive disease.
Time Frame: At 3 weeks (+/- 7 days) post Cycle 3 of the study treatment and prior to IDS.
Population: Participants who received any amount of assigned protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | DL1 Dose Escalation Cohort | DL1 Dose Expansion-only Cohort | DL2 Dose Escalation Cohort
Number analyzed (Participants) | 7 | 13 | 5
Participants
  Complete response | 0 | 1 | 0
  Partial response | 3 | 5 | 3
  Stable disease | 1 | 2 | 1
  Non-complete response/non-progressive disease | 2 | 3 | 0
  Progressive disease | 0 | 1 | 0
  Not evaluable | 1 | 1 | 1

5. Other Pre Specified Outcome: Phosphorylated (p)PRAS40 Expression in Tumor
Description: Will be summarized by collection time point and dose level. Wilcoxon signed rank test will be used to explore the change of pPRAS40 expression in the pre-treatment versus on-treatment tumor in the patients who have been treated at the maximum tolerated dose and have evaluable biopsy specimen.
Time Frame: Up to 90 days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Measurements of Tissue and Blood Pharmacokinetics for Ipatasertib
Description: Descriptive statistics (e.g., mean, standard deviation) will be given for the ipatasertib pharmacokinetics measured in the tissue and blood. Graphs and non-linear model techniques will be used to describe and identify the maximum plasma concentration (Cmax) and the time to observed Cmax (Tmax) for ipatasertib whenever these are applied.
Time Frame: Up to day of surgery
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Tumor Response
Description: Assessed by RECIST 1.1, and measurements for genomic alterations in PI3K Pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1). Summary statistics (or graphs) for PTEN loss, genomic alterations in PI3K pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1), transcriptomic alterations in PI3K Pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1) will be given. The association of objective tumor response with each of these biomarkers will be explored by appropriate statistical methods, e.g., Spearman's rank correlation coefficient for ordinal or interval type of biomarker data, chi-squared test for nominal type of biomarker data.
Time Frame: Up to 90 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Tumor Response
Description: Assessed by RECIST 1.1, and measurements for transcriptomic alterations in PI3K Pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1). Summary statistics (or graphs) for PTEN loss, genomic alterations in PI3K pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1), transcriptomic alterations in PI3K Pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1) will be given. The association of objective tumor response with each of these biomarkers will be explored by appropriate statistical methods, e.g., Spearman's rank correlation coefficient for ordinal or interval type of biomarker data, chi-squared test for nominal type of biomarker data.
Time Frame: Up to 90 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Tumor Response
Description: Assessed by RECIST 1.1, and measurement for PTEN loss. Summary statistics (or graphs) for PTEN loss, genomic alterations in PI3K pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1), transcriptomic alterations in PI3K Pathway genes (PTEN, PI3KCA, PIK3R1, AKT1, p53 loss, KRAS, NF1, TSC1/TSC1) will be given. The association of objective tumor response with each of these biomarkers will be explored by appropriate statistical methods, e.g., Spearman's rank correlation coefficient for ordinal or interval type of biomarker data, chi-squared test for nominal type of biomarker data.
Time Frame: Up to 90 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During treatment period and up to 90 days after the last dose of ipatasertib. The median for duration of study treatment was 68 days with a range from 1 day to 90 days.
Description: Participants who received any amount of protocol therapy.
Arm/Group | DL1 Dose Escalation Cohort | DL1 Dose Expansion-only Cohort | DL2 Dose Escalation Cohort
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 3/13 | 5/5
Other Adverse Events (participants affected / at risk) | 7/7 | 13/13 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DL1 Dose Escalation Cohort (N=7) | DL1 Dose Expansion-only Cohort (N=13) | DL2 Dose Escalation Cohort (N=5)
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Death Nos (General disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Thromboembolic Event (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DL1 Dose Escalation Cohort (N=7) | DL1 Dose Expansion-only Cohort (N=13) | DL2 Dose Escalation Cohort (N=5)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 4 | 3 | 5
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 2 | 1
Chest Pain - Cardiac (Cardiac disorders) | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1
Heart Failure (Cardiac disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 4 | 6 | 5
Constipation (Gastrointestinal disorders) | 3 | 5 | 3
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2 | 4
Stomach Pain (Gastrointestinal disorders) | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Belching (Gastrointestinal disorders) | 1 | 0 | 0
Pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1
Fever (General disorders) | 1 | 1 | 1
General Disorders And Administration Site Conditio (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 2 | 5 | 4
Gait Disturbance (General disorders) | 0 | 0 | 1
Edema Limbs (General disorders) | 2 | 0 | 1
Death Nos (General disorders) | 0 | 0 | 1
Allergic Reaction (Immune system disorders) | 2 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 3
Thrush (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1
Infections And Infestations - Other (Infections and infestations) | 0 | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 2 | 2
Weight Loss (Investigations) | 2 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 3
Neutrophil Count Decreased (Investigations) | 0 | 1 | 3
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 2
Inr Increased (Investigations) | 0 | 0 | 1
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 0 | 1
Electrocardiogram Qt Corrected Interval Prolonged (Investigations) | 0 | 0 | 1
Ejection Fraction Decreased (Investigations) | 0 | 0 | 1
Creatinine Increased (Investigations) | 1 | 0 | 0
Cholesterol High (Investigations) | 2 | 0 | 1
Cardiac Troponin T Increased (Investigations) | 0 | 0 | 2
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1
White Blood Cell Decreased (Investigations) | 1 | 1 | 3
Blood Bicarbonate Decreased (Investigations) | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 3 | 1 | 1
Alkaline Phosphatase Increased (Investigations) | 0 | 3 | 1
Alanine Aminotransferase Increased (Investigations) | 3 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 3
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Syncope (Nervous system disorders) | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1 | 2
Nervous System Disorders - Other (Nervous system disorders) | 0 | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 3 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Concentration Impairment (Nervous system disorders) | 0 | 1 | 0
Renal And Urinary Disorders - Other (Renal and urinary disorders) | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary Urgency (Renal and urinary disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 1 | 1
Glucosuria (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory, Thoracic And Mediastinal Disorders - (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Vascular Disorders - Other (Vascular disorders) | 0 | 0 | 1
Thromboembolic Event (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 2
Hypertension (Vascular disorders) | 0 | 1 | 2
Flushing (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT05276973/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT05276973/ICF_000.pdf